CLINICAL TRIAL: NCT05781425
Title: Neurofilament Light Chain as Biomarker for Bortezomib-induced Peripheral Neuropathy
Brief Title: Prediction of Getting Peripheral Neuropathy in Patients Treated With Bortezomib?
Acronym: NFL-BIOPAIN
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Sygehus Lillebaelt (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: AKF-401
Record Dates: First submitted 2023-02-15; First posted 2023-03-23 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Neurofilament light chain; NFL; Proteasome inhibitor; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Multiple Myeloma patients: Treatment naïve multiple myeloma patients. There is no intervention.

SUMMARY:
Investigation of which patients treated with bortezomib that have increased risk of developing peripheral neuropathy.

DETAILED DESCRIPTION:
The study aims to include 20 patients with multiple myeloma that are initiating bortezomib treatment. The patients must follow their normal treatment cycles while getting blood drawn during their treatment period however maximal 9 cycles.

Blood is dawn before treatment initiation and approximately once per cycle in order to measure neurofilament light chain (NFL) before and during treatment. The primary outcome is to relate the level of NFL during treatment with the level at baseline and as a secondary outcome to relate the level of NFL to the cumulative dose of bortezomib.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Must speak and understand Danish
* Must be able to and willing to give informed consent
* Diagnosed with myeloma and in need for treatment
* Must not be a candidate for transplantation and must be a candidate for bortezomib treatment.
* Must not previously have been treated with proteasome inhibitors
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) ≤ 3

Exclusion Criteria:

* Other underlying cancer disease - with exception of a) basal cell carcinoma, b) healed carcinoma in situ cervicis uteri, c) other cancer disease with minimal risk of recurrence or d) prostate cancer with low glean score
* Previous treatment with neurotoxic chemotherapy
* Known polyneuropathy or at diagnosis have polyneuropathy degree 1 with pain or degree 2 without pain.
* Simultaneous amyloidosis/POEMS syndrome
* Patients who have received chemotherapy previously and patients with diabetes, HIV and neurodegenerative diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Must be at least 18 years of age, must understand and speak Danish, must have multiple myeloma and be a candidate for treatment with bortezomib and must not be at candidate for cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Level of plasma neurofilament light chain | Baseline (before treatment initiation)
  Plasma neurofilament light chain before treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Between day 8 and 15 in cycle 1 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib.
Level of plasma neurofilament light chain | Day 1 in cycle 2 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 3 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 4 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 5 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 6 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 7 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 8 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).
Level of plasma neurofilament light chain | Day 1 in cycle 9 (each cycle is often between 3-6 weeks)
  Plasma neurofilament light chain during treatment with bortezomib. (Cycle length can vary).

SECONDARY OUTCOMES:
Level of plasma neurofilament relative to cumulative dose of bortezomib | From cycle 1 (each cycle is often between 3-6 weeks) and forward, maximum 9 cycles in total. An average of 1 year.
  Plasma neurofilament light chain relative to the cumulative dose of bortezomib in patients.
Degree of peripheral neuropathy | From cycle 1 (each cycle is often between 3-6 weeks) and forward, maximum 9 cycles in total. An average of 1 year.
  Using questionnaire Chemotherapy-induced peripheral neuropathy 20 (CIPN20), grading
Degree of peripheral neuropathy | From cycle 1 (each cycle is often between 3-6 weeks) and forward, maximum 9 cycles in total. An average of 1 year.
  Using Common Terminology Criteria for Adverse Events (CTCAE) version 5, grading 1-5 with 1 being the mildest case and 5 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Per Damkier, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Blood Diseases - Aarhus University Hospital, Aarhus
  - Department of Hematology - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No
Individual participant data cannot be shared due to general data protection regulation (GDPR).